CLINICAL TRIAL: NCT00902772
Title: A Single-Centre, Single-Dose, Double-Blind, Randomized, Placebo- and Active-Controlled Crossover Study to Evaluate the AbusePotential of AZD7325 in Healthy Recreational CNS Depressant Users
Brief Title: Study to Evaluate the Abuse Potential of AZD7325 in Healthy Recreational Central Nervous System (CNS) Depressant Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: D1140C00008
Record Dates: First submitted 2009-05-12; First posted 2009-05-15 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Recreational CNS Depressant Use
Keywords: Recreational CNS depressant; Abuse liability; Abuse potential; Healthy Recreational CNS Depressant Users
MeSH Terms: interventions — Lorazepam; 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- A (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- B (Active Comparator): Lorazepam
  Interventions: Drug: Lorazepam
- C (Active Comparator): Lorazepam
  Interventions: Drug: Lorazepam
- D (Active Comparator): Lorazepam
  Interventions: Drug: Lorazepam
- E (Experimental): AZD7325
  Interventions: Drug: AZD7325
- F (Experimental): AZD7325
  Interventions: Drug: AZD7325
- G (Experimental): AZD7325
  Interventions: Drug: AZD7325

INTERVENTIONS:
Drug: Lorazepam — mg, oral dose
  Arms: B; C; D
Drug: AZD7325 — mg, oral dose
  Arms: E; F; G
Drug: Placebo
  Arms: A

SUMMARY:
The purpose of this study is to examine the abuse potential of AZD7325.

ELIGIBILITY:
Inclusion Criteria:

* Recreational CNS depressant use, defined as at least 10 lifetime occasions of non-medical use of drugs with depressant/sedative properties and at least 1 non-medical use in the year prior to screening
* Body mass index (BMI) within the range of 19.0 to 33.0 kg/m2, inclusive, and a minimum weight of 50.0 kg at screening
* Willing and able to abide by all study requirements and restrictions

Exclusion Criteria:

* Unwillingness of inability to abstain from recreational drug use for the duration of the study from screening until follow-up
* Positive breath alcohol test prior to dosing
* Clinically significant abnormalities on physical examination, medical history, 12-lead ECG, vital signs, or safety laboratories

Ages: 18 Months to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-05; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scales | Daily during Visit 2 through 9

SECONDARY OUTCOMES:
Columbia Suicide-Severity Rating Scale | Prior to each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Myroslava K Romach, MD, Principal Investigator — Kendle Early Stage - Toronto
Locations (1):
- Research Site, Toronto, Ontario, Canada